CLINICAL TRIAL: NCT02957019
Title: A Phase I/II Study of the Tumor-targeting Human L19-IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Rituximab in Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow progression due to difficulties in finding eligible patients. Competitive clinical trials with innovative agents and new approved products leaddefinitive stop.
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2RTX-01/14
Record Dates: First submitted 2016-10-27; First posted 2016-11-07 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L19-IL2 + RTX (Experimental): Phase I (Dose definition):
  Cohorts of 3-6 patients will receive Rituximab on day 1 and 8 of the first 3-weeks cycle (C1D1 and C1D8, respectively) and on day 1 of the second 3-weeks cycle (C2D1). During two uninterrupted 3-weeks cycles, L19-IL2 will be administered on C1D1, C1D8, C1D15 and C2D1, C2D8, C2D15.
  Phase II (Activity Evaluation):
  During Phase II, 14 patients will receive Rituximab on C1D1 and C1D8 and on C2D1. Two uninterrupted 3-weeks cycles of L19-IL2 at the RD determined during Phase I will be administered on C1D1, C1D8 and C1D15 and C2D1, C2D8 and C2D15.
  Interventions: Drug: L19-IL2 - Ph I; Drug: L19-IL2 at RD - Ph II; Drug: Rituximab

INTERVENTIONS:
Drug: L19-IL2 - Ph I — Patients will receive increasing doses of L19-IL2 (0.32, 0.43, 0.57 and 0.76 Mio IU/kg of IL-2 equivalents per administration) during Phase I study
Drug: L19-IL2 at RD - Ph II — Patients will receive L19-IL2 at the RD defined during the Phase I part of the study
Drug: Rituximab — Patients will receive a fixed dose of Rituximab (375 mg/m2) per administration during Phase I and Phase II of the study

SUMMARY:
Phase I/II, open-label, multicenter, prospective study.

DETAILED DESCRIPTION:
Phase I - Dose definition: A prospective, open-label, multi-center Phase I dose escalation study in which cohorts of 3-6 patients will receive escalating doses of L19-IL2 in combination with a fixed dose of Rituximab (375 mg/m2).

Phase II - Activity Evaluation: Open-label, multi-center, prospective study during which 14 enrolled patients will receive a fixed dose of Rituximab (375 mg/m2) in combination with L19-IL2 at the RD defined during the Phase I part of the study.

The study is designed to establish whether L19-IL2, administered in combination with Rituximab is well tolerated and can achieve objective responses and clinical benefit to patients with relapsed or refractory DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD 20-positive DLBCL
* Patients must have experienced relapse after or not have achieved CR with standard R-CHOP-like treatment and must be ineligible for autologous stem cell transplantation or must have relapsed/progressed after autologous or allogeneic stem cell transplantation. In this last case, time lapse between autologous stem cell transplantation and beginning of L19-IL2 treatment must not be less than 4 weeks; in case of allogeneic stem cell transplantation, L19-IL2 treatment can start 4 weeks after removal of immunosuppressive drug(s).
* Presence of measurable lesions according to Revised response criteria for malignant lymphoma
* Males or females, age ≥ 18 years
* ECOG performance status ≤ 2
* Life expectancy of at least 12 weeks
* Absolute neutrophil count > 1.5 x 109/L
* Hemoglobin > 8.0 g/dL
* Platelets > 50 x 109/L
* Total bilirubin ≤ 30 µmol/L (or ≤ 2.0 mg/dl)
* No abnormal electrocardiogram findings requiring treatment
* ALT and AST ≤ 3.0 x the upper limit of normal range (ULN) (5.0 x ULN for patients with hepatic involvement with lymphoma)
* Serum creatinine < 2 x ULN
* Negative tuberculosis test (e.g. Quantiferon-assay)
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) Grade ≤ 1 unless otherwise specified above
* Negative serum pregnancy test (for women of child-bearing potential only) at screening
* If of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug
* Able to provide written Informed Consent
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Evidence of central nervous system lymphoma
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, Tis & Ti) or any cancer curatively treated < 5 years prior to study entry
* Hypersensitivity to Rituximab or to murine proteins, or to any of its excipients (Sodium citrate, Polysorbate 80, Sodium chloride, Sodium hydroxide, Hydrochloric acid)
* History of HIV infection or infectious hepatitis B or C
* Presence of active, severe infections (e.g., tuberculosis, sepsis and opportunistic infections or any infection requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study. Patients with a history of recurring or chronic infections or with underlying conditions which may further predispose them to serious infections should be excluded from the study.
* Active graft-versus-host disease in patients with a history of allogeneic stem cell transplantation
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris
* Inadequately controlled cardiac arrhythmias including atrial fibrillation
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria)
* Uncontrolled hypertension
* Ischemic peripheral vascular disease (Grade IIb-IV)
* Severe diabetic retinopathy
* Active autoimmune disease
* History of solid organ allograft
* Recovery from major trauma including surgery within 4 weeks prior to administration of study treatment
* Known history of allergy to IL2 or other human proteins/peptides/antibodies
* Positive serum pregnancy test (for women of child-bearing potential only) at screening
* Breast feeding female
* Anti-tumor therapy within 4 weeks of the administration of study treatment (except small surgery)
* Patient requires or is taking corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterionAny conditions that in the opinion of the investigator could hamper compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events that are related to treatment and classified as DLTs for each administered dosage - phase I study | Up to Day 21 of the Cycle 1 (cycle of 21 days)
  To assess the dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended dose (RD) of L19-IL2 in combination with Rituximab
The rate of patients with complete response CR after 2 cycles of treatment - phase II study | From Day 38 to Day 42

SECONDARY OUTCOMES:
The overall response rate (ORR) - phase I study | Up to 24 months
Median progression free survival (PFS) - phase I study | Up to 24 months
Median overall survival (OS) - phase I study | Up to 24 months
Pharmacokinetics assessment of L19-IL2 through blood sampling - phase I study | At Day 2 of Cycle 1
Human anti-fusion protein antibodies (HAFA) levels - phase I study | (1) at Day 2, (2) at Day 23, (3) from Day 38 to Day 42, (4) from Day 80 to Day 84
Percentage of Participants With On-Study Adverse Events (AEs) and Serious Adverse Events (SAEs) - phase II study | Up to 24 months
Percentage of Participants With Worst On-Study Hematological and Chemistry Abnormalities - phase II study | Up to 24 months
Number of Patients With Abnormal Physical Examinations - phase II study | Up to 24 months
Relative percentage difference in vital signs from baseline - phase II study | Up to 24 months
The overall response rate (ORR) - phase II study | Up to 24 months
Median progression free survival (PFS) - phase II study | Up to 24 months
Median overall survival (OS) - phase II study | Up to 24 months
Human anti-fusion protein antibodies (HAFA) levels - phase II study | (1) at Day 2, (2) at Day 23, (3) from Day 38 to Day 42, (4) from Day 80 to Day 84

CONTACTS AND LOCATIONS:
Locations (1):
- Münster University Hospital, Münster, Germany